CLINICAL TRIAL: NCT06484205
Title: Promoting Human Rights in Mental Health: Evaluation of the Effectiveness of the World Health Organization QualityRights Training in Italy Among Caregivers of People With Psychosocial Disabilities
Brief Title: Evaluation of the Effectiveness of the World Health Organization QualityRights Training in Italy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Mauro Giovanni Carta, Principal Investigator, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Verbale n39
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Caregiver Burden
Keywords: psychosocial disabilities; caregivers; online training
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: This is a Randomized controlled clinical trial with four evaluation times (T0 pre- treatment; T1 post treatment; T2 3 months after T1 and T2 6 months after T1; aimed at evaluating the effectiveness of the World Health Organization QualityRights training compared to a control intervention (another online training program) in improving caregivers' human rights knowledge and attitudes towards people with psychosocial disabilities as rights holders.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WHO QualityRights e-training (Experimental): Participants assigned to the intervention group (n 40) will participate in the WHO QualityRights (QR) online training course on "Mental Health, Recovery and Community Inclusion". The QR training aims to increase knowledge of the rights of people with psychosocial disabilities and to change negative attitudes towards them and their role as rights holders.
  Interventions: Other: WHO QualityRights e-training
- Emotional intelligence e-training (Active Comparator): Participants assigned to the control group (n 40) will receive the online "Emotional Intelligence Training for Informal Caregivers" offered by PeerCare.
  Interventions: Other: Emotional intelligence e-training

INTERVENTIONS:
Other: WHO QualityRights e-training — WHO QualityRights training provides the necessary skills to support people with psychosocial disabilities in advocating for their rights. The QualityRights online course includes six main modules: 1) Human Rights; 2) Human rights, mental health and disability; 3) Legal capacity and the right to decide; 4) Stop coercion, violence and mistreatment; 5) Quality services and inclusion in the community; 6) Mental health, well-being and recovery and it will take approximately 8 hours for completion. QualityRights course modules can be completed at each participant's pace and needs. The training is considered concluded once the quizzes provided at the end of each of the six modules have been successfully completed and upon completion of the course it will be possible to download your official WHO certificate from the QR platform.
  Arms: WHO QualityRights e-training
Other: Emotional intelligence e-training — This course offers caregivers resources and knowledge so that they are able to manage their emotions and gain quality in the care they provide to others and in their own lives. The course duration is similar to that of the QualityRights online course and is intended for caregivers of people with disabilities and others interested
  Arms: Emotional intelligence e-training

SUMMARY:
The research aims to promote human rights of people with psychosocial disabilities. The design will be a randomized controlled trial (RCT) with two groups. The intervention will consist of participation in an online training, with a central focus on the human rights of people with psychosocial disabilities. The measured outcomes will be knowledge of human rights, caregivers' attitudes towards people with psychosocial disabilities as rights holders, caregiver burden, depressive symptoms, and quality of life.

DETAILED DESCRIPTION:
Throughout the world, people with psychosocial disabilities are frequently exposed to human rights violations, such as discrimination and exclusion from society, inability to access health services, physical, sexual and psychological abuse, violence, neglect and denial of the right to legal capacity.

Another obstacle to access to care, to social inclusion and which encourages violations of the human rights of people with psychosocial disabilities is represented by the stigma and discrimination it entails.

Furthermore, caregivers themselves can also be the recipients of stigma, and previous research suggests it affects more than half of them.

This stigmatization represents a real burden, especially in emotional terms, for caregivers and can reduce access to support, resources and opportunities in the social sphere with an impact that also has repercussions on the person with psychosocial disabilities for whom they take care. treatment.

The importance of providing positive support to caregivers in their supporting role emerges; an increasingly broad evidence base underlines the benefits of caregiver involvement on the well-being of their family member, in particular it is associated with an improvement in the quality of life, a reduction in symptoms, the risk of relapses and hospital admissions.

In this context, Internet-based interventions can be a useful tool to increase the knowledge of caregivers of people with psychosocial disabilities and to reduce the physical and psychological consequences resulting from burden and stigma.

The implementation of a mental health human rights literacy intervention among caregivers is of crucial importance in the current context. This type of initiative aims to provide caregivers with the knowledge and skills needed to understand, respect, defend and promote the human rights of people with psychosocial disabilities and can help caregivers identify situations where the rights of people with psychosocial disabilities could be violated. Such action can contribute to the empowerment of caregivers and people with mental health conditions and can help combat the stigma and discrimination associated with mental disorders.

The specific objective of the research is to conduct a randomized controlled trial in Italy to evaluate the effectiveness of the World Health Organization QualityRights training compared to a control intervention (another online training program) in improving human rights knowledge and caregivers' attitudes towards people with psychosocial disabilities as rights holders.

ELIGIBILITY:
Inclusion Criteria:

* people aged 18 or over;
* caregivers of people with psychosocial disabilities relating to local mental health services;
* italian speaking people

Exclusion Criteria:

* individuals under 18 years of age;
* people who have already participated in the WHO QualityRights online course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-06-26 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Improving the knowledge about human rights and the attitudes of caregivers towards people with psychosocial disabilities | T0 (0 month), T1 (post intervention), T2; (3 months after post-intervention), T3 (6 months after post-intervention)
  To evaluate it will be used: the World Health Organization's Knowledge about the Rights of persons with psychosocial disabilities questionnaire (16 items). It was developed by World Health Organization (WHO) to assess knowledge about the rights included in the United Nations Convention on the Rights of Persons with Disabilities (UN CRPD), and The World Health Organization's questionnaire on the attitudes towards people with psychosocial disabilities as rights-holders (17 items). It was developed by WHO and includes three sub-scales: attitudes towards institutionalization and living independently in the community; attitudes toward mandatory treatment and coercion; attitudes toward people with psychosocial disabilities as decision-makers.

SECONDARY OUTCOMES:
Change from Baseline to post intervention and to follow-ups of The Short Form Health Survey (Quality of life) | T0 (0 month), T1 (post intervention), T2; (3 months after post-intervention), T3 (6 months after post-intervention)
  To evaluate it will be used: The Short Form Health Survey (SF-12), a brief version of SF-36 questionnaire, made up of twelve questions, values range from 12 to 47, includes the following dimensions: physical activity, disturbance in physical health, physical condition, self-assessment of health status, vitality, social activity and mental health assessed on a monthly basis . Higher scores recorded a greeting and better Quality of life
Change from Baseline to post intervention and to follow-ups of Patient Health Questionnaire-9 (Depressive symptoms) | T0 (0 month), T1 (post intervention), T2; (3 months after post-intervention), T3 (6 months after post-intervention)
  To evaluate it will be used: Patient Health Questionnaire-9 (PHQ-9) a short self-administered tool, values range from 0 to 27, used for screening, diagnosis, monitoring and measuring the severity of depression. It's composed of 9 items that correspond to the symptoms of major depression according to Diagnostic and statistical manual of mental disorders (DSM-IV) on last two weeks. Higher scores identify a greater presence of depressive symptoms.
Change from Baseline to post intervention and to follow-ups of Zarit Burden interview | T0 (0 month), T1 (post intervention), T2; (3 months after post-intervention), T3 (6 months after post-intervention)
  To evaluate it will be used: The Zarit Burden interview, a questionnaire for assessing the consequences that the care burden of a family member with chronic disabilities has on the caregiver. It is a self-assessment tool made up of 22 items with responses rated on a 5-point Likert scale: from 0 (never) to 4 (almost always) based on the degree of agreement with the individual items. The items investigate how the patient's disability impacts the caregiver's quality of life, psychological suffering, sense of guilt, financial difficulties, shame and social and family difficulties.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Cagliari, Cagliari, Italy